CLINICAL TRIAL: NCT02608203
Title: Impact of [68 Ga]-DOTANOC PET-CT on the Management of Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs): Prospective, Multicentric Study.
Brief Title: [68 Ga]-DOTANOC PET/CT in GEP-NETs
Acronym: GEP-NOC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-46; RCAPHM14_0345 (Registry Identifier: AP-HM)
Record Dates: First submitted 2015-11-09; First posted 2015-11-18 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors

ARMS (1):
- patients with gastroenteropancreatic neuroendocrine tumors (Experimental)
  Interventions: Drug: [68Ga]-DOTANOC PET/CT

INTERVENTIONS:
Drug: [68Ga]-DOTANOC PET/CT

SUMMARY:
Somatostatin receptors are overexpressed in GEP-NETs and can be visualized in vivo by radiolabeled somatostatin-analogs.

During the last decades, conventional scintigraphy using 111In-DTPA-Octreotide (often named somatostatin receptor scintigraphy or SRS) was considered as the gold standard nuclear imaging technique in the evaluation of GEP-NETs. However, SRS may be suboptimal in this clinical setting because of the low intrinsic resolution of the technique and its selectivity for SST2 only. Its overall sensitivity is estimated to 60-70% (per lesion analysis), even when using the most recent SPECT-CT cameras. MRI have also a higher sensitivity than CT and SRS for the detection of liver metastases from GEP-NETs.

In recent years, positron emission tomography (PET) imaging, a high resolution and sensitive technology, has gained an increasing role in oncology. It has also been evaluated in GEP-NETs with somatostatin agonists (SSTa) radiolabelled with Gallium-68 [68Ga], a positron emitter with very promising results. Its diagnostic sensitivity is clearly superior to SRS and many European centers have already replaced SRS by [68Ga]-PET-SSTa.

Currently, three different [68Ga]-coupled peptides can be used in trials: DOTA-TOC, DOTA-TATE and DOTA-NOC with excellent affinities for SST2 (IC50: 2.5; 0.2 and 1.9 nM, respectively). Sensitivities of DOTA-TOC and DOTA-TATE PET/CT are quite similar.

[68Ga]-DOTANOC which also binds to SST5 was recently found to detect significantly more lesions than the SST2-specific radiotracer [68Ga]-DOTATATE in patients with GEP-NETs but this requires further evaluation.

It is therefore important to determine the interest of [68Ga]-DOTANOC combined with the standard diagnosis strategy in GEP-NETs and evaluate medicoeconomic impact of adding [68Ga]-DOTANOC in the work-up of patients.

The investigators hypothesis is that [68Ga]-DOTANOC will modify the management in at least 20% of patients in a more adapted way according to the 2012 ENETS guidelines in comparison to the decision based on the standard imaging work up (multiphasic WB CT, liver MRI and SRS).

110 patients will be included prospectively in 5 different French experienced centers (Marseille, Bordeaux, Toulouse, Paris, Clermond-Ferrand).

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18 years, with affiliation to the Social Security.
2. Written consent of the patient.
3. Patients with any of the following 5 situations:

   * GEPs without metastasis.
   * GEPs with unilateral liver metastases candidates to unilateral hepatectomy.
   * GEPs with unknown primary tumor.
   * GEPS with livers metastases candidates to liver transplantation.
   * Metastatic GEPs with grade 1 or 2 tumour and negative SRS.
4. Reference imaging within the last 3 months : multiphasic total body CT scan, liver MRI and SRS (SPECT/CT).

Exclusion Criteria:

1. minor subject.
2. Pregnant or breast-feeding.
3. Absence of therapeutic alternatives in metastatic GEP.
4. Undifferentiated GEP and/or metastatic GEPs with grade 3 tumours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
level of changes (%) between care management before DOTANOC PET and care management after DOTANOC PET | 6 months

SECONDARY OUTCOMES:
Positive predictive values of DOTANOC PET and standard imaging | 1 year
negative predictive values of DOTANOC PET and standard imaging | 1 year
correlation between tumor type and DOTANOC PET results | 1 year
number of patients for whom PET allowed the detection of lesions not described by standard imaging | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — AP-HM
Locations (1):
- AP-HM, Marseille, France